CLINICAL TRIAL: NCT02122614
Title: The Role of Home-monitoring in the Adherence of Patients With Chronic Obstructive Pulmonary Disease to Long-term Rehabilitation
Brief Title: Home-monitoring and Adherence of Patients With COPD to Long-term Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SFRH/BD/81328/2011
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; COPD; Pulmonary rehabilitation; Physical activity; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: Pulmonary rehabilitation (PR) plus PA monitoring and feedback from a pedometer
- Control group (Active Comparator)
  Interventions: Behavioral: Pulmonary rehabilitation (PR)

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation (PR) plus PA monitoring and feedback from a pedometer — Patients will enrol in a 12-week PR program comprising exercise training (3 times per week) and psychoeducation sessions (once a week). Patients will also receive a pedometer to self-monitor their PA during and after the PR program and individualized step-count goals.
  Arms: Experimental group
Behavioral: Pulmonary rehabilitation (PR) — Patients will enrol in a 12-week PR program comprising exercise training (3 times per week) and psychoeducation sessions (once a week).
  Arms: Control group

SUMMARY:
The aim of this randomized controlled trial is to investigate the effects of adding PA monitoring and regular feedback of a pedometer (step counter) to an outpatient pulmonary rehabilitation (PR) program on daily PA levels and health status of patients with COPD.

Patients will be randomized to either receive a PR program with PA monitoring and regular feedback of a pedometer (experimental group [EG]) or a PR program alone (control group [CG]). During the PR program, patients in the EG will receive a pedometer to self-monitor their PA and individualized step-count goals. They will continue to use the pedometers and receive individualized goals for 3 months after the program.

It is expected that, by receiving individualized goals and a simple pedometer to self-monitor their PA during and after a PR program, patients with COPD will become more active and adhere to long-term rehabilitation, thus reducing the overall impact of COPD.

DETAILED DESCRIPTION:
Patients with Chronic Obstructive Pulmonary Disease (COPD) present lower levels of physical activity (PA), which have been associated with increased healthcare utilization and reduced survival. Thus, optimizing PA levels has become one therapeutic priority in COPD management.

Pulmonary rehabilitation (PR) is an effective intervention in reducing symptoms and improving patients' functional status and quality of life. However, its effects in increasing patients' physical activity (PA) levels are limited. Previous research has suggested that PR with continuous PA monitoring with feedback may be a suitable approach to increase and maintain patients' PA levels.

Patients who agree to participate will be randomized to either receive a PR program with PA monitoring and regular feedback of a pedometer (experimental group [EG]) or a PR program alone (control group [CG]). Both PR programs will last 12 weeks and consist of exercise training and psychoeducation sessions. During the PR program, patients in the EG will receive a pedometer to self-monitor their PA and individualized step-count goals. They will continue to use the pedometers and receive individualized goals for 3 months after the program.

The impact of the intervention will be explored using a mixed-methods approach.

Assessments will be conducted in both groups at 4 time points: before, immediately after, 3 and 6 months after the PR program. Physical activity levels, lung function, breathlessness, exercise tolerance, peripheral muscle strength, health-related quality of life and healthcare utilization will be assessed in both groups in these time points.

Descriptive statistics will be used to characterize the sample. To analyze changes in outcome measures, data from the two groups will be compared at each time point.

Patients in the EG will also be invited to attend focus groups after the intervention to assess their perspective about the intervention and their satisfaction with the use of the pedometer.

A sample size calculation using the primary outcome was performed based in a previous pilot study. It was found that 12 patients with COPD would be required in each group to provide 80% power (alpha = 0.05) to detect significant differences between groups. However, as PR programs usually have considerable dropouts (around 30%), 16 patients with COPD were recruited for each group.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria
* ≥ 18 years old
* clinical stability for 1 month prior to the study (no hospital admissions or exacerbations)
* able to provide their own informed consent

Exclusion Criteria:

* inability to understand and co-operate
* presence of severe psychiatric conditions
* presence of severe neurologic/ musculoskeletal conditions and/or unstable cardiovascular disease
* participation in regular strenuous exercise (e.g., greater than 10 hours per week of running, swimming, weightlifting or any other similar physical activity) prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity levels | 1 week before, 1 week after, 3 and 6 months after the PR program
  Physical activity data will be collected using a triaxial accelerometer. Number of steps per day and time spent in sedentary, light and moderate-to-vigorous intensity activities will be assessed. Time spent in different postures (i.e., standing, sitting and lying) will also be determined.

SECONDARY OUTCOMES:
Change in exercise tolerance | 1 week before, 1 week after, 3 and 6 months after the PR program
  Exercise tolerance will be assessed with the 6-minute walk test, following the American Thoracic Society guidelines. The maximal distance walked during 6 minutes and the associated respiratory symptoms will be collected.
Change in peripheral muscle strength | 1 week before, 1 week after, 3 and 6 months after the PR program
  Isometric muscle strength of the upper and lower limbs will be assessed with the 1 repetition maximum (1-RM), following the American College of Sports Medicine guidelines.
Change in activities limitation resulting from breathlessness | 1 week before, 1 week after, 3 and 6 months after the PR program
  The Modified British Medical Research Council questionnaire comprises five grades (statements) in a scale from 0 to 4, with higher grades indicating greater perceived respiratory limitation.
Change in behavioral regulations in exercise | 1 week before, 1 week after, 3 and 6 months after the PR program
  The Behavioural Regulation in Exercise Questionnaire-2 (BRES-2) is a 19-item instrument designed to measure different forms of motivation for physical exercise and includes 5 sub-scales.
Change in general self-efficacy | 1 week before, 1 week after, 3 and 6 months after the PR program
  The Self-Efficacy Scale is an instrument designed to measure general self-efficacy. Higher scores indicate higher self-efficacy.
Change in health-related quality of life | 1 week before, 1 week after, 3 and 6 months after the PR program
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure quality of life in patients with chronic lung disease. It has 3 domains: symptoms, activities and impact. Higher scores indicate poorer quality of life.
Patients' perspectives about the intervention (experimental group only) | Immediately after the intervention
  Semi-structured focus group interviews will be conducted with patients to explore the impact of the intervention (i.e., Pulmonary rehabilitation plus PA monitoring and feedback from a pedometer).

OTHER OUTCOMES:
Change in lung function | 1 week before, 1 week after, 3 and 6 months after the PR program
  Lung function will be assessed with spirometry, according to the American Thoracic Society/European Respiratory Society guidelines.
Change in the number and duration of respiratory exacerbations and hospitalizations | 1 week before, 1 week after, 3 and 6 months after the PR program
  The number and duration of respiratory exacerbations and hospitalizations will be assessed during patients' interview.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Aveiro District, Portugal

REFERENCES:
- [Background] Cruz J, Brooks D, Marques A. Home telemonitoring in COPD: a systematic review of methodologies and patients' adherence. Int J Med Inform. 2014 Apr;83(4):249-63. doi: 10.1016/j.ijmedinf.2014.01.008. Epub 2014 Jan 23. PMID 24529402
- [Background] Cruz J, Brooks D, Marques A. Home telemonitoring effectiveness in COPD: a systematic review. Int J Clin Pract. 2014 Mar;68(3):369-78. doi: 10.1111/ijcp.12345. Epub 2014 Jan 28. PMID 24472009
- [Background] Cruz J, Brooks D, Marques A. Impact of feedback on physical activity levels of individuals with chronic obstructive pulmonary disease during pulmonary rehabilitation: A feasibility study. Chron Respir Dis. 2014 Nov;11(4):191-8. doi: 10.1177/1479972314552280. Epub 2014 Oct 2. PMID 25278009
- [Derived] Cruz J, Brooks D, Marques A. Walk2Bactive: A randomised controlled trial of a physical activity-focused behavioural intervention beyond pulmonary rehabilitation in chronic obstructive pulmonary disease. Chron Respir Dis. 2016 Feb;13(1):57-66. doi: 10.1177/1479972315619574. Epub 2015 Dec 23. PMID 26703921